CLINICAL TRIAL: NCT05719896
Title: A Phase II, Double-blind, Randomized, Parallel-group, Placebo-controlled Trial to Evaluate the Efficacy and Safety of DT01 Tablets in Patients With Irritable Bowel Syndrome With Diarrhea
Brief Title: Efficacy and Safety of DT01 Tablets in Patients With Irritable Bowel Syndrome With Diarrhea
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre of Clinical Pharmacology, Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC001-1
Record Dates: First submitted 2022-12-10; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-12

CONDITIONS: Irritable Bowel Syndrome With Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo tablets (Placebo Comparator): Posology: oral administration of 3 placebo tablets three times per day for 8 weeks.
  Interventions: Drug: Placebo tablets
- DT01 tablets (Experimental): Posology: oral administration of 3 DT01 tablets three times per day for 8 weeks.
  Interventions: Drug: DT01 tablets
- DT01-Placebo tablets (Experimental): Posology: oral administration of 2 DT01 tablets and 1 placebo tablet, three times per day for 8 weeks.
  Interventions: Drug: DT01-Placebo tablets

INTERVENTIONS:
Drug: DT01 tablets — Each subject was given orally 3 DT01 tablets/day for 8 weeks
  Arms: DT01 tablets
Drug: Placebo tablets — Each subject was given orally 3 DT01 tablets/day for 8 weeks
  Arms: Placebo tablets
Drug: DT01-Placebo tablets — Each subject was given orally 2 DT01 tablets and 1 Placebo tablet, three times per day for 8 weeks
  Arms: DT01-Placebo tablets

SUMMARY:
This is a Phase II, double-blind, randomized, 3-arm, placebo-controlled study to evaluate the efficacy and describe the safety of DT01 tablets in adults with IBS-D.

Patients who meet all entry criteria will be randomized to receive DT tablets or placebo or both for 8 weeks. The study drug will be taken three times daily. Investigators will conduct phone-based assessments on Days 7, 14, 21, 28, 35, 42, 49. Patients will return to the clinic after dosing has completed (Day 56) for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Has a diagnosis of IBS-D (Irritable Bowel Syndrome with Diarrhea) and meets the Rome IV Criteria
* Additional criterion: more than 3 bowel movements per day at least 25% of the time in the last 3 months.
* For patients older than 50 years OR patients with a positive family history of colorectal cancer: Normal results from colonoscopy/flexible sigmoidoscopy performed within the last 2 years.
* For patients aged 65 years or older: Absence of ischaemic colitis, microscopy colitis or any other organic gastrointestinal disease as evidenced by the results of a colonoscopy/flexible sigmoidoscopy with biopsy performed within 12 months.
* Mentally competent, able to give written informed consent, and compliant to undergo all visits and procedures.
* Unrestricted access to a touch-tone telephone.
* Willingness to refrain from using loperamide within 3 days prior to run-in visit and during the run-in period.
* For women of childbearing potential: Use of a highly effective contraceptive method with a failure rate <1% per year throughout the entire study period.

Additional criteria at randomisation: During both weeks of the run-in period:

1. A weekly average of worst abdominal pain in the past 24 hours with a score of ≥ 3.0 according to the Visual Analogue Scale (VAS).
2. At least one bowel movement on each day.
3. A weekly average of at least 3 bowel movements per day.
4. At least one stool with a consistency of Type 6 or Type 7 according to the Bristol Stool Scale (BSS) on at least 2 days per week.
5. Less than 2 bowel movements with a consistency of Type 1 or Type 2 according to the BSS per week.
6. Adequate compliance with the diary recording procedure defined as at least ≥80% of the nominal daily data entry.

Exclusion Criteria:

* Diagnosis of IBS with a subtype of constipation, mixed IBS, or un-subtyped IBS.
* History of organic GI abnormalities, inflammatory bowel diseases, complicated diverticulosis, ischaemic colitis, microscopic colitis.
* History of pancreatitis, active biliary duct disease, cholecystitis or symptomatic gallbladder stone disease in the previous 6 months.
* History of gluten enteropathy or lactose intolerance.
* Hypersensitivity to the active substances or to any of the excipients of study drug or placebo.
* History of major cardiovascular events in the previous 6 months.
* History of human immunodeficiency virus infection.
* Uncontrolled hypertension, insulin-dependent diabetes mellitus or abnormal thyroid function.
* Evidence of clinically significant hepatic disease, severe renal insufficiency or anemia.
* Use of prohibited concurrent medication within the previous month such as antibiotics, antimuscarinic drugs, drugs enhancing GI motility and analgesics.
* Pregnancy or breastfeeding.
* Inability to understand or collaborate throughout the study.
* Participation in other clinical studies in the previous 4 weeks or concomitant enrollment in a clinical study.
* Any condition that would compromise the well-being of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Abdominal pain response | 8 weeks
  Decrease in the weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline
Stool consistency response | 8 weeks
  Decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 according to the Bristol Stool Scale (BSS) compared with baseline.
Weekly response for abdominal pain intensity and stool consistency over 8 weeks of treatment in at least 50% of the weeks of treatment (4 out of 8 weeks) | 8 weeks
  A participant must meet both of the Abdominal pain response and Stool consistency response in the same week to be a weekly responder.

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Traditional Medicine, Hanoi, Vietnam